CLINICAL TRIAL: NCT05695001
Title: An Open Observational Prospective Pilot Study of the Efficacy and Safety of Cytokine Hemosorption Using the Efferon CT Device in Acute Endogenous Intoxication in Patients With Acute Pancreatitis and Aseptic Pancreatic Necrosis
Brief Title: Hemoperfusion Efferon СT for the Treatment of Patients With Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Other Study IDs: efferon-ct-2022-02
Record Dates: First submitted 2023-01-13; First posted 2023-01-23 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Acute Pancreatitis With Uninfected Necrosis, Unspecified
Keywords: acute pancreatitis; sepsis; cytokine sorption; endogenous intoxication
MeSH Terms: conditions — Pancreatitis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No Intervention: Baseline therapy: Basic therapy is the routine practice of an institution for the treatment of patients with acute pancreatitis without signs of infection
- Experimental: Basic therapy + Efferon CT: Basic therapy is a routine practice of the institution for the treatment of patients with acute uninfected pancreatitis in combination with extracorporeal hemoperfusion (Efferon CT)
  Interventions: Device: Efferon CT

INTERVENTIONS:
Device: Efferon CT — Efferon CT is a cylindrical body made of polycarbonate, filled with spherical granules of polymer hemocompatible macroporous styrene-divinylbenzene copolymer of super cross-linked type and isotonic sodium chloride solution. The device is manufactured according to TU 32.50.50-001-12264678-2018, has passed the necessary tests and is registered in Russia as a medical product RZN 2019/8886.
  Groups: Experimental: Basic therapy + Efferon CT

SUMMARY:
Mortality from severe acute pancreatitis reaches 42%. The prognosis of acute pancreatitis is associated with the development of acute inflammatory response syndrome (SIRS) and multiple organ failure (MOF). Due to the lack of etiological therapy, the treatment of acute pancreatitis is predominantly symptomatic.

Severity and mortality are associated with early systemic inflammatory response syndrome (SIRS) and septic complications at a later stage of the disease.

With regard to the pronounced inflammatory response ("cytokine storm") during the early phase of endogenous intoxication of acute pancreatitis, extracorporeal removal of cytokines is a promising therapeutic approach.

This prospective study examines the effect of early extracorporeal sorption of cytokines using the Efferon CT device on the severity of clinical symptoms of endogenous intoxication in acute pancreatitis and aseptic pancreatic necrosis.

DETAILED DESCRIPTION:
Acute pancreatitis in emergency surgery takes the 3rd place in terms of the frequency of its manifestation, second only to acute appendicitis and cholecystitis. The incidence of acute pancreatitis is growing from year to year and is more than 38 patients per 10,000 population per year. In 25% of patients, the development of pancreatitis is destructive.

Mortality in this pathology is mainly associated with the development of severe necrotic forms that cause a systemic inflammatory response of the body. The formation of pancreatic necrosis occurs within 1-2 days of illness, and it is at this time that the therapeutic effect is most effective. Quite often, upon admission of a patient, the severity of his condition, the data of laboratory and instrumental methods of examination do not allow us to judge the further course of the disease.

The existing systems and scales for assessing the severity of the patient APACHE II, SAPS, MODS, SOFA, Glasgow, J. Ranson and others provide an acceptable accuracy of about 80% only after 48 hours from the onset of the disease, and before that time they are of little information. This means that the severity of the condition of 20% of patients with necrotizing pancreatitis cannot be assessed in time by these systems until its clinical deterioration is obvious. Thus, often, the time when adequate treatment can affect the outcome of the disease is missed. After that, against the background of the picture of pancreatic necrosis, complications arise at lightning speed and like an avalanche, despite the measures taken to prevent them.

In this regard, the earliest identification of patients with an aggressive, destructive nature of the disease for the entire complex of intensive care seems to be very important. The severity of the patient's condition with acute pancreatitis is largely determined by the severity of endotoxemia. The latter, in turn, depends on the cytokine response of the body. "Cytokine storm", which occurs in the acute phase of pancreatitis, leads to aggravation of intoxication, inadequate and untimely correction of which underlies the development of pancreatogenic shock, multiple organ failure and septic complications.

To date, the early pathogenetic mechanisms of acute pancreatitis and its complications are poorly understood. The question of what happens at the subcellular level, what processes are responsible for the development of severe forms of the disease, extraorganic complications remains insufficiently studied.

Treatment of acute pancreatitis is traditionally divided into conservative and surgical. The start time of conservative measures, their components, an adequate assessment of effectiveness affect the timing and extent of surgical intervention.

At the moment, there is no specific surgical tactics for sterile and infected pancreatic necrosis, as well as for its purulent-septic complications. It is known that lethality from infected pancreatic necrosis is 2-3 times higher than from a sterile process.

The severity of the patient's condition with acute pancreatitis is largely determined by the severity of endotoxemia. The latter, in turn, depends on the cytokine response of the body.

In connection with the increasing spread of the "cytokine theory" in the past 10 years, various methods of extracorporeal detoxification have become widespread in the practice of intensive care for severe forms of acute pancreatitis. Despite this, there is no consensus among specialists regarding the timing of the application of certain techniques in the context of the phase course of acute pancreatitis, the required frequency of procedures, and their effectiveness.

In acute pancreatitis, severe endotoxemia occurs early, which leads to the development of multiple organ failure. Allocate biochemical, immunological and microbial components of endogenous intoxication, which include intermediate and final metabolites of the processes of autolysis and secondary infection.

Detoxification underlies the prevention and pathogenetic treatment of complications of acute pancreatitis. Numerous tests have shown that the use of extracorporeal sorption methods, the eliminirinducing pro-inflammatory cytokines, improves the results of treatment of patients with manifestations of endogenous intoxication.

Many techniques have been described - hemofiltration (HF), enterosorption, ultrahemofiltration (UHF), hemosorption (HS), plasmapheresis (PF). Very few studies have been devoted to the use of the hemosorption method in the early stage of development of acute pancreatitis, before the appearance of septic complications.

Recently, there has been a search for new approaches to the treatment of patients in the early stages of pancreatitis, even before the development of formidable complications, significantly worsening the prognosis of the disease. One of them may be extracorporeal removal from the systemic circulation of excessively produced mediators of the inflammatory response (cytokines) by hemosorption.

Hemosorption is the most modern method of removing substances toxic to body cells from the patient's blood. The procedure is carried out outside the body by pumping the blood flow through a column filled with a sorbent (hemoperfusion procedure). Critical parameters for therapeutic efficacy are the type of sorbent, its volume, the number of repeated procedures; they are individualized depending on the identified pathological disorders and the patient's condition.

Currently, there are no multicenter randomized studies confirming the need for extracorporeal blood purification methods as one of the main areas of pathogenetic therapy for acute pancreatitis. At the same time, the increasing emergence of data on the significant influence of the "cytokine storm" on the pathogenesis of the disease and its progressive deterioration suggests a possible positive role of the cytokine hemosorption method performed in the early phase of acute pancreatitis.

Efferon CT (JSC Efferon, Moscow, Russia) is a device for extracorporeal blood purification using direct hemoperfusion. Detoxification is carried out by sorption of cytokines and other products of endogenous intoxication with a molecular size of up to 55 kDa.

In connection with the above data, the purpose of this clinical study is to determine the degree of influence of the use of the hemosorption device Efferon CT (JSC Efferon, Russia) on the clinical manifestations and laboratory parameters of acute pancreatitis occurring without septic complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old,
* Verified diagnosis of "Acute pancreatitis" according to the Atlanta classification of acute pancreatitis (2012), without signs of infection,
* No more than 72 hours from the onset of an attack of acute pancreatitis to hemosorption,
* The patient's condition allows for therapy with the Efferon CT device for at least 4 hours.

Exclusion Criteria:

* History of chronic pancreatitis (exacerbation of chronic pancreatitis),
* The presence of a focus of non-sanitized surgical infection,
* The use of other methods of extracorporeal removal of inflammatory mediators in the treatment of pancreatitis (hemofilters with highly permeable and surface-modified membranes),
* Inability to achieve or maintain a minimum mean arterial pressure (MAP) ≥ 65 mmHg. Art., despite vasopressor therapy and infusion therapy for 24 hours,
* End-stage renal disease, and the need for chronic dialysis,
* Acute pulmonary embolism,
* Transfusion reaction,
* Severe congestive heart failure,
* The patient has had an acute myocardial infarction within the last 4 weeks,
* Uncontrolled bleeding (acute blood loss in the last 24 hours),
* Severe granulocytopenia (white blood cell count less than 500 cells/mm3) or severe thrombocytopenia,
* Oncopathology out of remission.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes over 18 years of age with signs of acute pancreatitis no later than 72 hours from the onset of an attack of pain without signs of an infectious process
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Effect of Efferon CT hemoperfusion on SOFA scores (Sequential Organ Failure Assessment) in patients with acute pancreatitis. | 1-72 hours
  The value of indicators on the SOFA scale every 24 hours ± 1 hour from the start of hemoperfusion (0 hour) to 72 hours. The SOFA index is equal to the sum of six indicators. The higher the score, the greater the insufficiency of the system being assessed. The higher the overall index, the greater the degree of multiorgan dysfunction. Violation of the function of each organ (system) is assessed separately in dynamics against the background of intensive therapy. With a score of no more than 12, multiple organ dysfunctions are assumed, 13-17 points indicate the transition of dysfunction to insufficiency, a score of about 24 indicates a high probability of death. The lower the SOFA index, the less pronounced organ failure and the better the patient's survival prognosis.

SECONDARY OUTCOMES:
The effect of Efferon CT hemoperfusion on length of stay in the intensive care unit | 1-14 days
  Time (number of days) from enrollment in the study to transfer from the intensive care unit within 14 days.
Effect of Efferon hemoperfusion on interleukin levels (IL-1b, IL-6, IL-8, IL-10, IL-18) | 1-72 hours
  The significance of interleukin levels before the start of hemoperfusion and 72 hours after the start of hemoperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kiselev, PhD, MD, Principal Investigator — N. V. Sklifosovsky Moscow Research Institute of Emergency, Moscow, Russia
Locations (1):
- N.V. Sklifosovsky Moscow Research Institute of Emergency, Moscow, Russia